CLINICAL TRIAL: NCT04540081
Title: Enhancing Electronic Health Systems to Decrease the Burden of Colon Cancer, Lung Cancer, Obesity, Vaccine-Preventable Illness, and LivER Cancer
Acronym: CLOVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1624888
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2021-11

CONDITIONS: Colon Cancer; Lung Cancer; Tobacco Use Cessation; Obesity; Pneumonia, Bacterial; Shingles; Hepatitis C
MeSH Terms: conditions — Colonic Neoplasms; Lung Neoplasms; Tobacco Use Cessation; Obesity; Pneumonia, Bacterial; Herpes Zoster; Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLOVER arm (Experimental): This arm will contain clinics that utilize the CLOVER intervention
  Interventions: Other: Epic Healthy Planet Population Health Module
- Standard of Care arm (No Intervention): This arm will contain clinics that do not utilize the CLOVER intervention

INTERVENTIONS:
Other: Epic Healthy Planet Population Health Module — Electronic population health module which is tailored to increased adherence to USPSTF and CDC recommendations
  Arms: CLOVER arm

SUMMARY:
The purpose of CLOVER is to utilize Epic Healthy Planet to increase adherence to United States Preventive Services Task Force (USPSTF) and Centers for Disease Control and Prevention (CDC) recommendations in adults age 50 and older.

ELIGIBILITY:
Inclusion Criteria:

- Any patient who has a UC Davis or UC Irvine primary care provider (PCP) and is deficient in any of the following: colon cancer screening, lung cancer screening, tobacco cessation counseling, obesity counseling, pneumonia vaccination, shingles vaccine, and hepatitis C screening.

Exclusion Criteria:

- Patients outside of the age limits or have an established PCP.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20000 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Overall Adherence to CLOVER Metrics | 6 months
  This is the proportion of patients who appropriately completed screenings and vaccinations that they were eligible for

SECONDARY OUTCOMES:
Colon cancer screening | 6 months
  Proportion of eligible patients who completed colon cancer screening.
Lung cancer screening | 6 months
  Proportion of eligible patients who completed lung cancer screening.
Tobacco cessation counseling | 6 months
  Proportion of eligible patients who completed tobacco cessation counseling.
Obesity counseling | 6 months
  Proportion of eligible patients who completed obesity counseling.
Pneumonia vaccination | 6 months
  Proportion of eligible patients who completed pneumonia vaccination.
Shingles vaccination | 6 months
  Proportion of eligible patients who completed shingles vaccination.
Hepatitis C screening | 6 months
  Proportion of eligible patients who completed hepatitis C screening.

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided